CLINICAL TRIAL: NCT05326685
Title: The Effect of Visual Video With Korotkoff Sounds on Blood Pressure Measurement Skills and Anxiety Levels: A Randomized Controlled Study
Brief Title: The Effect of Visual Video With Korotkoff Sounds on Blood Pressure Measurement Skills and Anxiety Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Turkan Ulker, MSc, RN, Research Asistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 31
Record Dates: First submitted 2022-04-01; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Anxiety
Keywords: Anxiety; Blood Pressure Measurement Skills; Korotkoff sounds; Nursing students
MeSH Terms: conditions — Anxiety Disorders | interventions — Videotape Recording

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): video with korotkoff sounds
  Interventions: Other: video with korotkoff sounds
- Control (No Intervention): standart practice

INTERVENTIONS:
Other: video with korotkoff sounds — The State-Trait Anxiety Inventory short version (STAIS-5, STAIT-5) and the student introduction form were applied at the beginning of the study. Then Intervention participants were shown and listened visual video with korotkoff sounds before blood presssure measurement. Afterwards, blood pressure was measured to the students 3 times and 3 measurements were recorded. After the application about 2 hours later, the students State Anxiety Inventory short version (STAIS-5) form was filled again by students.
  Arms: Intervention

SUMMARY:
Background: The aim of this study was to determine the effect of visual video with korotkoff sounds on nursing students' blood presssure measurement skills and anxiety levels.

Methods: This was a randomized controlled experimental study conducted at the nursing department of the faculty of health sciences of a university. Intervention participants were shown and listened visual video with korotkoff sounds before blood presssure measurement. Aural and visual video containing Korotkoff sounds were shown to the students before the practice.

DETAILED DESCRIPTION:
Background: The aim of this study was to determine the effect of visual video with korotkoff sounds on nursing students' blood presssure measurement skills and anxiety levels.

Methods: This was a randomized controlled experimental study conducted at the nursing department of the faculty of health sciences of a university. Intervention participants were shown and listened visual video with korotkoff sounds before blood presssure measurement. Aural and visual video containing Korotkoff sounds were shown to the students before the practice. The data of the research were collected with the State-Trait Anxiety Inventory short version (STAIS-5, STAIT-5) and the Student introduction form.

ELIGIBILITY:
Inclusion Criteria:

* Studying in the first year of the nursing department in the 2021-2022 academic year,
* Taking the "pulse and blood pressure measurement" course and laboratory practice
* Students who agree to participate in the study will be included.

Exclusion Criteria:

* Previous manual blood pressure measurement experience,
* Those who do not participate in the theoretical part of the "pulse and blood pressure measurement" course,
* Students who do not attend the lesson on the day of the applications will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-03-11 (Actual); Study Completion 2022-03-27 (Actual)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory (STAIS-5, STAIT-5) | pre intervention
  State-Trait Anxiety Inventory short version (STAIS-5, STAIT-5)[ Time Frame: pre-intervention ] The STAI consists of two parts; the State Anxiety Inventory (SAI) and the Trait Anxiety Inventory (TAI). The SAI measures anxiety about an event while the TAI measures anxiety level as a personal characteristic. The STAIS-5, STAIT-5 each consists of 5 items. The scale items are scored on a 4-point Likert scale of 0 to 3 (0= Not at all, 1= Somewhat, 2= Moderately so, 3= Very much so). Higher scores indicate greater anxiety. The scale allow researchers to differentiate among anxious and healthy participants.

SECONDARY OUTCOMES:
State Anxiety Inventory (STAIS-5) | through study completion for each group, an average of 2 hours
  The SAI items are scored on scored on a 4-point Likert scale of 0 to 3 (0= Not at all, 1= Somewhat, 2= Moderately so, 3= Very much so). Higher scores indicate greater anxiety
Practice Success | through study completion for each participant, an average of 2 hours
  blood pressure was measured to all students 3 times and all measurements were recorded. the instructors informed students about BPM and then paired them up, who then took each other's blood pressure using a sphygmomanometer and a stethoscope with headphones that enable both the participant and the instructors to listen to Korotkoff sounds. The instructors evaluated the participants'BPM performanceby listening to the Korotkoff sounds by one of the headphones and by monitoring the manometer

CONTACTS AND LOCATIONS:
Overall Officials: TÜRKAN ÜLKER, Principal Investigator — TC Erciyes University
Locations (1):
- Türkan Ülker, Kayseri, Turkey (Türkiye)